CLINICAL TRIAL: NCT03511495
Title: Repeatability and Reliability of Galilei Corneal Topographer Measurements in Keratoconus
Brief Title: Reliability of Topography Measurements in Keratoconus
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Assistant Professor of Ophthalmology, Milton S. Hershey Medical Center
Other Study IDs: STUDY00007951
Record Dates: First submitted 2018-03-28; First posted 2018-04-27 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Keratoconic Patients
  Interventions: Diagnostic Test: Galilei Corneal Topographer

INTERVENTIONS:
Diagnostic Test: Galilei Corneal Topographer — A series of five measurements via the Galilei corneal topographer of each keratoconic eye in quick succession

SUMMARY:
The purpose of this study is to assess the reliability and repeatability of the parameters obtained using the Galilei dual-scheimpflug corneal topographer for monitoring progression in eyes with keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a progressive corneal degeneration characterized by progressive steepening and thinning of the central or paracentral cornea leading to corneal protrusion and resulting irregular astigmatism and high myopia. This disorder is usually bilateral and is linked to atopy and excessive eye rubbing, although the precise pathophysiology behind development of this condition is unclear. Keratoconus is the most common corneal degeneration in the United States, affecting between 50 and 230 subjects per 100,000 population.

Early diagnosis and appropriate management of keratoconus relies greatly on accurate assessment of corneal topographic measurements. It is therefore imperative that the data obtained via corneal topography devices is accurate and reliable.

The GALILEI Dual Scheimpflug Analyzer integrates Placido disc topography and dual Scheimpflug tomography to assess anterior and posterior corneal curvature data. Although there have been several studies performed assessing the ability of the Galilei to accurately distinguish keratoconus from unaffected eyes and investigating interdevice reliability between the Galilei analyzer and other tomographers, to our knowledge the repeatability of measurements obtained in this population via the Galilei device has been incompletely evaluated to date.

Corneal topography data obtained via the Galilei device is relied upon heavily in clinical decision making for keratoconic patients both in the Hershey Eye Clinic and in a great number of ophthalmology practices world-wide. It is vital that the accuracy and repeatability of these measurements obtained via the Galilei device are investigated.

The primary endpoint to be measured in the study will be the maximum (steepest) and minimum (flattest) keratometry values in the central zone.

Secondary endpoints will be maximum keratometry across the entire area scanned, axis of corneal astigmatism, anterior and posterior best fit spheres in float mode with the diameter set to 8 mm, maximum anterior and posterior elevations, thinnest corneal thickness, and corneal asphericity at 6 mm, root mean square (RMS) of the HOAs, RMS of the third-order coma, coma axis, vertical and horizontal coma and spherical aberration.

ELIGIBILITY:
Inclusion Criteria:

* Patientswho are older than 18 years of age
* Patients who are scheduled to undergo Galilei dual-scheimpflug corneal topography testing
* Patients who have been diagnosed with keratoconus
* Measurements with a reported reliability of 'good' from the topographer

Exclusion Criteria:

* Patients who have undergone any prior surgical intervention involving the cornea (i.e. cornea transplant or INTACS, or corneal cross linking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study of patients seen at the Penn State Eye Center who have been diagnosed with keratoconus and are undergoing Galilei corneal topography. Patients will be selected to participate in the study based on inclusion/exclusion criteria. Each patient in the study will undergo five consecutive corneal topography measurements per keratoconic eye.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum (steepest) and minimum (flattest) keratometry values in the central zone | Measured at day 0 of study enrollment
  Assessment of the steepness of the cornea

SECONDARY OUTCOMES:
Thinnest pachymetry | Measured at day 0 of study enrollment
  The thinnest area of the cornea

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pantanelli, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Eye Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Bawazeer AM, Hodge WG, Lorimer B. Atopy and keratoconus: a multivariate analysis. Br J Ophthalmol. 2000 Aug;84(8):834-6. doi: 10.1136/bjo.84.8.834. PMID 10906086
- [Background] Demir S, Sonmez B, Yeter V, Ortak H. Comparison of normal and keratoconic corneas by Galilei Dual-Scheimpflug Analyzer. Cont Lens Anterior Eye. 2013 Oct;36(5):219-25. doi: 10.1016/j.clae.2013.04.001. Epub 2013 Apr 30. PMID 23642799
- [Background] Holladay JT. Keratoconus detection using corneal topography. J Refract Surg. 2009 Oct;25(10 Suppl):S958-62. doi: 10.3928/1081597X-20090915-11. PMID 19848378
- [Background] Guler E, Yagci R, Akyol M, Arslanyilmaz Z, Balci M, Hepsen IF. Repeatability and reproducibility of Galilei measurements in normal keratoconic and postrefractive corneas. Cont Lens Anterior Eye. 2014 Oct;37(5):331-6. doi: 10.1016/j.clae.2014.04.004. Epub 2014 Jun 14. PMID 24938125
- [Background] Meyer JJ, Gokul A, Vellara HR, Prime Z, McGhee CN. Repeatability and Agreement of Orbscan II, Pentacam HR, and Galilei Tomography Systems in Corneas With Keratoconus. Am J Ophthalmol. 2017 Mar;175:122-128. doi: 10.1016/j.ajo.2016.12.003. Epub 2016 Dec 18. PMID 27993593
- [Background] Feizi S, Yaseri M, Kheiri B. Predictive Ability of Galilei to Distinguish Subclinical Keratoconus and Keratoconus from Normal Corneas. J Ophthalmic Vis Res. 2016 Jan-Mar;11(1):8-16. doi: 10.4103/2008-322X.180707. PMID 27195079
- [Background] Jahadi Hosseini HR, Katbab A, Khalili MR, Abtahi MB. Comparison of corneal thickness measurements using Galilei, HR Pentacam, and ultrasound. Cornea. 2010 Oct;29(10):1091-5. doi: 10.1097/ICO.0b013e3181cf98e5. PMID 20628301
- [Background] Anayol MA, Guler E, Yagci R, Sekeroglu MA, Ylmazoglu M, Trhs H, Kulak AE, Ylmazbas P. Comparison of central corneal thickness, thinnest corneal thickness, anterior chamber depth, and simulated keratometry using galilei, Pentacam, and Sirius devices. Cornea. 2014 Jun;33(6):582-6. doi: 10.1097/ICO.0000000000000119. PMID 24763122
- [Background] Park SH, Choi SK, Lee D, Jun EJ, Kim JH. Corneal thickness measurement using Orbscan, Pentacam, Galilei, and ultrasound in normal and post-femtosecond laser in situ keratomileusis eyes. Cornea. 2012 Sep;31(9):978-82. doi: 10.1097/ICO.0b013e31823d03fc. PMID 22699561
- [Background] Crawford AZ, Patel DV, McGhee CN. Comparison and repeatability of keratometric and corneal power measurements obtained by Orbscan II, Pentacam, and Galilei corneal tomography systems. Am J Ophthalmol. 2013 Jul;156(1):53-60. doi: 10.1016/j.ajo.2013.01.029. Epub 2013 Mar 28. PMID 23540708